CLINICAL TRIAL: NCT02132663
Title: The Effects on Growth and Tolerance of a Routine Infant Formula Fed to Term Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mead Johnson Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 3386-1
Record Dates: First submitted 2014-05-05; First posted 2014-05-07 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Growth of Term Infants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Infant formula containing an alternate source of DHA (Experimental)
  Interventions: Other: An investigational infant formula containing an alternate source of DHA
- Marketed routine infant formula (Active Comparator)
  Interventions: Other: Control: Marketed routine infant formula

INTERVENTIONS:
Other: Control: Marketed routine infant formula
  Arms: Marketed routine infant formula
Other: An investigational infant formula containing an alternate source of DHA
  Arms: Infant formula containing an alternate source of DHA

SUMMARY:
This clinical trial will evaluate an investigational infant formula with an alternate source of DHA to determine if it provides normal growth and if it is well tolerated by term infants as compared to a marketed routine infant formula.

ELIGIBILITY:
Inclusion Criteria:

* Singleton, 10-14 days of age at randomization
* Term infant with birth weight of a minimum of 2500 grams
* Solely formula fed
* Signed Informed Consent and Protected Health Information

Exclusion Criteria:

* History of underlying metabolic or chronic disease or immunocompromised
* Feeding difficulties or formula intolerance

Ages: 10 Days to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 315 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Body weight measured at each study visit | 3.5 Months

SECONDARY OUTCOMES:
Recall of infant formula intake at each study visit | 3.5 months
Body length measured at each study visit | 3.5 months
Recall of stool consistency measured at each study visit | 3.5 months
Medically-confirmed adverse events collected throughout the study period | 3.5 months
Head circumference measured at each study visit | 3.5 months
Recall of gastrointestinal tolerance measured at each study visit | 3.5 months
Blood Collection | Once at 120 days of age
  Blood Collection from a subset of participants to measure levels of fatty acids such as docosahexaenoic acid (DHA) and arachidonic acid (ARA).

CONTACTS AND LOCATIONS:
Overall Officials: Carol Lynn Berseth, M.D., Study Director — Mead Johnson and Company
Locations (22):
- United States (22):
  - Birmingham Pediatric Associates, Birmingham, Alabama
  - Greenvale Pediatrics - Hoover, Birmingham, Alabama
  - Southeastern Pediatric Association, Dothan, Alabama
  - Pediatrics East - Alabama Clinical Therapeutics, Pinson, Alabama
  - Northwest Arkansas Pediatric Clinic, Fayetteville, Arkansas
  - The Children's Clinic of Jonesboro, P.A., Jonesboro, Arkansas
  - Norwich Pediatric Group, PC, Norwich, Connecticut
  - Children's Research, LLC, Altamonte Springs, Florida
  - Physician Care Clinical Research, Sarasota, Florida
  - Deaconess Clinical Research, Evansville, Indiana
  - Owensboro Pediatrics, Owensboro, Kentucky
  - Woburn Pediatic Associates, Woburn, Massachusetts
  - Cary Pediatric Center, Cary, North Carolina
  - Capital Pediatrics & Adolescent Center, Raleigh, North Carolina
  - Pediatric Associates of Mt. Carmel, Inc, Cincinnati, Ohio
  - Pediatric Associates of Fairfield, Inc., Fairfield, Ohio
  - UHMP Comprehensive Pediatrics, Westlake, Ohio
  - Coastal Pediatric Research, Charleston, South Carolina
  - The Jackson Clinic - North Jackson, Jackson, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Austin Diagnostic Clinic, Austin, Texas
  - DCOL Center for Clinical Research, Longview, Texas

REFERENCES:
- [Derived] Yeiser M, Harris CL, Kirchoff AL, Patterson AC, Wampler JL, Zissman EN, Berseth CL. Growth and tolerance of infants fed formula with a new algal source of docosahexaenoic acid: Double-blind, randomized, controlled trial. Prostaglandins Leukot Essent Fatty Acids. 2016 Dec;115:89-96. doi: 10.1016/j.plefa.2016.09.001. Epub 2016 Sep 29. PMID 27914519